CLINICAL TRIAL: NCT03134950
Title: Improving Care for Youth With Functional Abdominal Pain: A Stepped Care Cognitive Behavioral Therapy (CBT) Delivery Approach
Brief Title: Improving Care for Youth With FAP: A Stepped Care CBT Delivery Approach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michigan State University (Other)
Collaborators: American Pain Society (Other); Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Principal Investigator, Natoshia Cunningham, Assistant Professor, Michigan State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-1388
Record Dates: First submitted 2017-04-12; First posted 2017-05-01 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Functional Abdominal Pain Syndrome; Anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — Analgesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ADAPT (Experimental): Aim to Decrease Anxiety and Pain Treatment (ADAPT) is a tailored CBT ranging from 4 sessions (pain-focused) to 6 sessions (blend of pain and anxiety coping strategies depending on the needs of the individual patients. The first 2 sessions are in person with a trained psychologist and the following 2-4 sessions are web-based. Each web-based session is followed by phone support.
  Interventions: Behavioral: ADAPT
- Medical Treatment as Usual (No Intervention): Medical treatment as usual

INTERVENTIONS:
Behavioral: ADAPT — Aim to Decrease Anxiety and Pain Treatment is a tailored CBT ranging from 4 sessions (pain-focused) to 6 sessions (blend of pain and anxiety coping strategies depending on the needs of the individual patients. The first 2 sessions will be in person with a trained psychologist and the following 2-4 sessions will be web-based. Each web-based session will be followed by phone support.
  Other Names: Aim to Decrease Anxiety and Pain Treatment
  Arms: ADAPT

SUMMARY:
This project aims to test a stepped care behavioral intervention approach for youth with functional abdominal pain (FAP) that is feasible to administer in medical settings. Screening and a brief intervention (i.e. psychoeducation and relaxation training) are provided to youth with FAP with more than minimal functional disability (FDI score >7) during their medical visit as part of enhanced usual care (EUC). Patients are re-assessed after two weeks. Those that fail to respond to EUC (as evidenced by FDI score >7) are eligible to undergo a baseline assessment and then are randomized to receive either 1) a more intensive and tailored CBT approach, Aim to Decrease Anxiety and Pain Treatment (ADAPT), provided by a trained psychologist, or 2) medical treatment as usual (TAU). It is hypothesized that youth who participate in ADAPT will have lower average pain rating scores, less pain-related functional disability, and less anxiety symptoms (if elevated) at post-assessment as compared to youth receiving medical TAU.

DETAILED DESCRIPTION:
The goal of this project is to pilot test different levels of behavioral intervention for patients diagnosed with FAP who are presenting for pediatric gastroenterology care. Patients are screened during their medical visit. Those with more than minimal levels of functional disability (Functional Disability Inventory (FDI) score >7), receive Enhanced Usual Care (EUC), brief pain-focused psychoeducation administered as part of their medical visit. As part of EUC, patients receive access to a web module for home use that reiterates educational material and offers relaxation training tools for home practice (i.e., audio recordings). Two weeks following EUC, patient outcomes are re-assessed with a focus on pain-related disability. Those who fail to respond to EUC (i.e., FDI remains >7) are invited to complete the next phase of the study. Eligible participants undergo a baseline assessment consisting of a diagnostic interview and child measures pertaining to pain, anxiety, depressive symptoms, and pain-related worries. Caregivers complete forms about their child's pain history, child disability, and child worries. Caregivers also complete a form about their own stress symptoms. After baseline assessment, patients are randomized to medical treatment as usual (TAU) or ADAPT, a tailored CBT delivered by a trained psychologist. ADAPT content differs based on the individual needs of the patient (i.e., all patients receive 4 pain-focused coping skills sessions, and those who present with clinical levels of anxiety receive 2 additional sessions to address anxiety symptoms). Participants complete 4 or 6 sessions (2 in person sessions and 2-4 web modules with phone support). Approximately six weeks after randomization, the patient and caregiver undergo follow-up assessment to assess pain, anxiety, and disability. It is hypothesized that youth who participate in ADAPT will have lower average pain rating scores, less pain-related functional disability, and lower levels of anxiety symptoms (if elevated) at post-assessment as compared to youth receiving medical TAU.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with functional abdominal pain by a pediatric gastroenterologist
* clinically significant disability evidenced by a total score of > 7 on the Functional Disability Inventory (FDI) that remains elevated (>2) after 2 weeks

Exclusion Criteria:

* significant medical condition(s) with an identifiable organic cause (e.g., Inflammatory Bowel Diseases such as Ulcerative Colitis and Chron's Disease)
* documented developmental delay, severe cognitive impairment, or a thought disorder
* evidence of severe depressive symptoms (CDI 2: T score >80) and/or active suicidal ideation

Ages: 9 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 139 (Actual)
Dates: Start 2015-07-20 (Actual); Primary Completion 2018-02-08 (Actual); Study Completion 2018-02-08 (Actual)

PRIMARY OUTCOMES:
Functional Disability Inventory - Child Version (FDI-C) | through study completion, an average of 8 weeks
  A 15-item self report inventory measuring perceived pain-related disability

SECONDARY OUTCOMES:
Screen for Child Anxiety Related Disorders - Child Report (SCARED-C) | through study completion, an average of 8 weeks
  Patient-reported measure of anxiety symptoms over the past 3 months
Pain Intensity via a Visual Analog Scale (VAS) | through study completion, an average of 8 weeks
  Average pain levels in the past 2 weeks using a 0 -10 scale
Anxiety Disorder Interview Schedule - Child Version (ADIS) | through study completion, an average of 8 weeks
  A validated interview conducted by a clinician to assess for childhood psychiatric disorders, with a focus on anxiety
Child Depression Inventory 2 Self Report (CDI-2) | through study completion, an average of 8 weeks
  A self report inventory measuring symptoms of depression in children and adolescents.
Pain Catastrophizing Scale for Children, Child Version (PCS-C) | through study completion, an average of 8 weeks
  An adaptation of the Pain Catastrophizing Scale used to study coping styles among child chronic pain patients.
Functional Gastrointestinal Disorders (FGIDs) Questionnaire | through study completion, an average of 8 weeks
  This questionnaire is based off of the ROME III diagnostic criteria and is used to validate patients' FGID diagnosis. Administered by research staff.
Children's Somatization Inventory (CSI-24) | through study completion, an average of 8 weeks
  A questionnaire that assesses the perceived severity of 24 nonspecific somatic symptoms. Items are based off of the symptom criteria for somatization disorders as defined by the Diagnostic and Statistical Manual of Mental Disorders (DSM).
Depression Anxiety Stress Scales (DASS21) | through study completion, an average of 8 weeks
  A brief self-report measure to assess parent negative-emotional states of depression, anxiety, and tension/stress.
Children's Global Assessment Scale (C-GAS) | through study completion, an average of 8 weeks
  A 0-100 scale anchored with descriptors of the patient ranging from "extremely impaired" to "doing very well". The study clinician completes the C-GAS after the completion of the ADIS.
Affective Reactivity Index (ARI) | through study completion, an average of 8 weeks
  A validated measure of irritability in pediatric populations

CONTACTS AND LOCATIONS:
Overall Officials: Natoshia Cunningham, PhD, Principal Investigator — Michigan State University
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

REFERENCES:
- [Derived] Kalomiris AE, Ely SL, Love SC, Mara CA, Cunningham NR. Child-Focused Cognitive Behavioral Therapy for Pediatric Abdominal Pain Disorders Reduces Caregiver Anxiety in Randomized Clinical Trial. J Pain. 2022 May;23(5):810-821. doi: 10.1016/j.jpain.2021.12.001. Epub 2021 Dec 11. PMID 34902549
- [Derived] Cunningham NR, Kalomiris A, Peugh J, Farrell M, Pentiuk S, Mallon D, Le C, Moorman E, Fussner L, Dutta RA, Kashikar-Zuck S. Cognitive Behavior Therapy Tailored to Anxiety Symptoms Improves Pediatric Functional Abdominal Pain Outcomes: A Randomized Clinical Trial. J Pediatr. 2021 Mar;230:62-70.e3. doi: 10.1016/j.jpeds.2020.10.060. Epub 2020 Oct 31. PMID 33130153